CLINICAL TRIAL: NCT02004626
Title: Study Phase III, Randomized, Double-blind, Multicenter, National, to Evaluate the Non-inferiority in Efficacy of Investigational Product Regarding the Comparator Product, in Debridement of Devitalized Tissue in Uninfected Pressure Ulcers.
Brief Title: Evaluate the Noninferiority of Medicines Treating Uninfected Pressure Ulcers.
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Cristália Produtos Químicos Farmacêuticos Ltda. (Industry)
Collaborators: Newco Trials Pesquisa Científica Ltda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRT071
Record Dates: First submitted 2013-10-28; First posted 2013-12-09 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Pressure Ulcer
Keywords: Collagenase; Phase III; National; Noninferiority; Double-blind; Multicenter; Prospective.
MeSH Terms: conditions — Pressure Ulcer | interventions — Collagenases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Collagenase (Active Comparator): Each gram of ointment contains :
  Collagenase ...0.6 U
  Vehicle qs ... 1 g
  Presentation:
  Topic use. 5 g tube of ointment containing smooth, lump-free , pale white to slightly brown with faint characteristic odor .
  Dosage The ointment should have full contact with the entire injured area, and uniformly applied twice a day.
  Interventions: Drug: Collagenase
- Kollagenase (Active Comparator): Each gram of ointment contains :
  Collagenase ... 0.6 U
  Vehicle qs ... 1 g
  Presentation
  Topic use. 5 g tube of ointment containing brownish clear, fat and weak characteristic odor.
  Dosage The ointment should have full contact with all the injured area, being uniformly applied twice a day.
  Interventions: Drug: Kollagenase

INTERVENTIONS:
Drug: Collagenase — Conduction of security tests: complete coagulation and glycosylated hemoglobin. Volunteers in childbearing age, with β-HCG (human chorionic gonadotropin) test.
  Verification of anthropometric data, clinical evaluation, PU evaluation, randomization and treatment start.
  Wash the wound with 0.9 % sterile saline solution; Apply of the investigational product directly in the devitalized tissue (necrotic tissue and Slough).
  Cover the wound with sterile gauze and dry transparent film. The procedures for the exchange of bandages must be done every day, twice a day until the total debridement of devitalized tissue.
  Photographic records.
  Arms: Collagenase
Drug: Kollagenase — Conduction of security tests: complete coagulation and glycosylated hemoglobin. Volunteers in childbearing age, with β-HCG (human chorionic gonadotropin) test.
  Verification of anthropometric data, clinical evaluation, PU evaluation, randomization and treatment start.
  Wash the wound with 0.9 % sterile saline solution; Apply of the investigational product directly in the devitalized tissue (necrotic tissue and Slough).
  Cover the wound with sterile gauze and dry transparent film. The procedures for the exchange of bandages must be done every day, twice a day until the total debridement of devitalized tissue.
  Photographic records.
  Arms: Kollagenase

SUMMARY:
This is a Clinical study Phase III, Prospective, Randomized, Controlled, Double-blind, Multicenter, National, Non-inferiority.

Its purpose is to determine the noninferiority in efficacy of an investigational product in relation to the product available in the market intended of treating pressure ulcers.

DETAILED DESCRIPTION:
Objectives:

The primary objective of efficacy is the reduction in the area of devitalized tissue based on the photographic record.

The secondary objective is to evaluate:

* formation of granulation tissue;
* the lesion reduction during treatment;
* the healing process of the Pressure Ulcer (PU) range of PUSH;
* the safety of the investigational product.

Study Plan:

* Estimated 92 research participants;
* Aged between ≥ 18 years and ≤ 80 years - both sexes;
* Visits from 1 to 10;
* The maximum lasting period in the study for each research participant will be approximately four weeks.

Evaluations During Study:

Evaluation of Digital Photography: The digital photographic record can provide the relative size of the wound, the tissue color and condition of the surrounding skin. The evaluation of digital photograph of each research participant will be performed by the classification assigned to the decrease of devitalized area and tissue e repair related to the time of healing and observed the formation of granulation tissue and epithelialization from standardized photographs.

Evaluation by PUSH Scales:

In order to provide an evaluation instrument of PUs in Brazil, so that satisfies the simplicity of the use in different clinical scenarios keeping its measurement properties, as previously attested from its original version, the PUSH scale was adapted into Portuguese.

The PUSH Scale considers three parameters or sub - scales of the wound healing process and treatment outcomes: wound area, amount of exudate present on the wound, appearance of the wound.

Retention of Records:

The investigator shall retain all documentation of the study over a period of at least five years from the end of the study. The Sponsor or its designee will provide a list of all documentation which should be kept by the Investigator.

Monitoring:

All aspects of the study will be carefully monitored by Cristália Pharmaceutical Chemicals Ltda. or designated representative of it (Clinical Research Organization - CRO) for evaluations related to good clinical practice and applicable local regulations.

Case Report Forms:

The Monitor will be available if the investigator, or other person of his team, needs information and guidance.

The Monitor of the study should have permanent access to all documentation and it is his obligation to ensure that the Case Report Forms are complete and completed correctly, as well as checking if the data are described according to the source documents, in order to eliminate interferences that may compromise the accuracy of the data generated in the clinical trial.

Audit and Inspections:

Authorized representatives of the Sponsor or designees, regulatory authority or the Ethics Committee of the institution may conduct audits or inspections during or after the study conclusion.

Collecting Data:

The information corresponding to the data of interest from the study will be collected and recorded in Case Report forms provided by Sponsor, and filled from the information contained in the source documents.

Documents are considered sources for study: medical records used by the professional at the time of the visits, diagnostic tests or image.

Informed Consent of Trial:

The Principal Investigator will ensure that the research participant receive verbally and in writing all relevant information about the nature, purpose, the test drug, the possible risks and benefits of the study.

Research participants will be notified that they are free to discontinue the study at any time. That they will have the opportunity to ask questions and to have sufficient time to consider the information received.

Formation of the database:

The database of the study will be assembled with the data from the Case Report Forms. Doubts and discrepancies will generate questions (queries) written to the Principal Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes;
* Aged ≥ 18 years and ≤ 80 years;
* Patients hospitalized;
* Patients with leg ulcers in the sacral region with presence of devitalized/ necrotic tissue indicating conservative debridement;
* Understanding, agreement and signing the Informed Consent Form (IFC), and the Authorization Term for the Image Use for publication of results

Exclusion Criteria:

* Infected ulcers;
* Limited ulcers;
* Ulcers with indication for surgical debridement ;
* Periostitis ;
* Obesity II( BMI ≥ 35 ) ;
* Severe malnutrition ( BMI < 16 )
* Hemoglobin (HbA1c ) above the upper limit of normal (ULN ) ;
* Coagulation Factor twice the ULN ;
* Patients with pulmonary emphysema and / or Chronic Obstructive Pulmonary Disease (COPD) ;
* Collagen diseases;
* Psychiatric illnesses;
* Patients using cytotoxic agents ;
* Oncology patients under palliative care ;
* Outpatients ;
* Signs of limb ischemia ;
* Urinary incontinence uncontrolled;
* Fecal incontinence;
* Diarrhea that in the opinion of the investigator , compromise the process of debridement;
* Known allergy from the components of the formulas;
* Pregnancy ;
* Breastfeeding ;
* Local and concomitant use of medications and / or products in the lesion: tyrothricin , gramicidin , tetracycline , hexachlorophene , heavy metals ( mercury, silver) , iodine , potassium permanganate , hydrogen peroxide , soap, detergent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Devitalized tissue reduction. | A month.
  Percentage of the area reduction of devitalized tissue, surrounding the injury total area and devitalized tissue for each 2D photographic record, with the use of standard metric, using the software IMAGE® J.

SECONDARY OUTCOMES:
Injury reduction. | A month.
  Evaluation of the wound area, related to the greatest length (in cephalo-caudal direction) versus the greatest width (horizontal line from right to left) in square centimeters, using the software IMAGE® J.
Granulation tissue formation. | A month.
  Classification assigned to the reduction of devitalized area and from tissue repair related to the time for healing and verified by formation of granulation and epithelialization tissue from standardized photographs using the software IMAGE® J.
Healing process of PU. | A month.
  Evolution of the healing process of PU by PUSH Scale.
Adverse events. | A month.
  Frequency and percentage of adverse effects occurrence by the participants of the research.

CONTACTS AND LOCATIONS:
Overall Officials: Norton Marcos S. Castro, Medic, Principal Investigator — Clínica Dr. Norton Sayeg Ltda
Locations (1):
- Clínica Dr. Norton Sayeg Ltda, São Paulo, São Paulo, Brazil